CLINICAL TRIAL: NCT05756036
Title: Torque Teno Virus: A Biomarker of Immunosuppression in Kidney Transplantation, an Observational Single Centre Study
Brief Title: Torque Teno Virus: A Biomarker of Immunosuppression
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 291391
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Renal Transplant Rejection; Immunosuppression; Renal Transplant Failure; Renal Transplant Infection
Keywords: renal transplant; immunosuppression; Torque teno virus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Renal transplant recipients: All incident renal transplant recipients after the commencement of the study
  Interventions: Other: None Observational study

INTERVENTIONS:
Other: None Observational study — Non interventional study

SUMMARY:
To seek an association between Torque Teno Virus DNA titres resulting from under or over-immunosuppression in a kidney allograft recipient, Graft rejection, both cell-mediated rejection and antibody-mediated rejection, donor-specific antibodies (DSA), the incidence of BK viraemia and BK nephropathy, CMV infection or diseases and PCP infection and the number of circulating NK, B and T lymphocyte subtypes.

DETAILED DESCRIPTION:
Balancing the adverse effects of over-immunosuppression such as infection and malignancy, to the risk of rejection, remains the central challenge for day-to-day clinical practice in transplantation. A quantitative measure of immunocompetence remains elusive, and in the absence of such markers, immunosuppression drug concentrations and clinical events, such as organ rejection, infection, malignancy etc. are used as surrogate markers of immunocompetence to guide therapy. As demonstrated in several studies, the Torque teno virus is widespread amongst the general population. In theory, if one suppresses the immune system, these viruses should multiply, resulting in a higher DNA level which can be detected by a simple blood test. Hence, the DNA level could be used as an indicator for the level of immunosuppression, along with the available blood tests to measure the level of toxicity of the said drugs.

In this research to be done at the Royal London Hospital, the investigators aim to elucidate that the Torque teno virus is widely prevalent in an ethnically diverse East London kidney transplant recipient population by conducting the viral PCR on blood samples already collected during their routine clinic visits. The population will include all kidney transplant recipients in a two-year period. The investigators will measure the correlation between the TTV DNA level and drug concentrations of the immunosuppressive medications which will elucidate how the DNA levels are affected by different drug concentrations. The investigators will then measure the correlation between the TTV DNA levels, and the common adverse outcomes experienced by the transplant recipients, namely, patient death, loss of transplant organs, transplant rejection, rates of infection, and cancers in transplant patients by collecting data from patient records. These tests will help understand whether the Torque teno virus DNA levels can be used as a marker of immunosuppression in the general population in the UK.

ELIGIBILITY:
Inclusion Criteria:

* All consenting renal transplant recipients in the study period will be included in the study

Exclusion Criteria:

* no exclusion criteria.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consenting renal transplant recipients in the study period
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The correlation between TTV viral load and Biopsy proven graft rejection | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No